CLINICAL TRIAL: NCT01436409
Title: Comparison of the Rates of Fetal Extractions Between a Systematic Practice of an Echography of Presentation and the Only Vaginal Touch Usually Realized During the Labor
Brief Title: Rates of Fetal Extractions Between Only Vaginal Touch Usually Realized and Vaginal Touch + Echography
Acronym: PINKFINGER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P050304; 2005/0570 (Other: DGS)
Record Dates: First submitted 2011-08-08; First posted 2011-09-19 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-07

CONDITIONS: Assisted Delivery
Keywords: vaginal touch; deliveries assisted; echography; assisted delivery
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- only vaginal touch (Other)
  Interventions: Other: echography
- vaginal touch +echography (Experimental)
  Interventions: Other: echography

INTERVENTIONS:
Other: echography — echography during labor

SUMMARY:
The main objective of this study is to compare the rate of fetal extractions between a systematic practice of an echography of presentation and the vaginal touch only one usually realized during the labor.

DETAILED DESCRIPTION:
The main objective is to compare the rate of fetal extractions between a systematic practice of an echography of presentation and the vaginal touch only one usually realized during the labor.

It is a prospective, randomized study. After randomization, the patients will be assigned to one of following both groups:

* Diagnosis of the variety of presentation of the fetal head by the usual examination, that is the only vaginal touch allowing the palpation of the sutures of the fetal head to locate the axis and the orientation of this one in the maternal pond. However, this clinical examination can be completed by an echography if the team considers that this information is necessary to optimize the coverage delivery in case of extraction by pair of forceps or suction cup.
* Diagnosis of the variety of presentation of the fetal head by the vaginal touch, confirmed by the systematic practice of an abdominal echography completed by a perineal echography from 8 cms of dilation, and made for a maximal extension of 15 minutes following the vaginal touch. This echography will be at the need repeated

  1900 patients (that is 950 by group) have to allow to detect a decrease of 25 % of the rate of deliveries assisted in the experimental group (systematic echography) with regard to the control group (TV), that is a decrease absolved from the rate from 20 % to 15 %, with a 80 % power and a risk of 5 % (bilateral test).

Duration of participation in the study: = 2 days Duration of the inclusions: 36 months

Criteria of efficiency Rate of deliveries attended defined by a composite criteria: deliveries by caesarian from a dilation of the cervix = 8 cms, and instrumental extractions by pair of forceps or suction cup.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* singleton pregnancy in head presentation
* gestational age ≥ 37 WG
* dilation of the cervix = 8 cms

Exclusion Criteria:

* caesarian antecedent, preeclampsia, praevia placental
* maternal and pregnancy pathology
* included in other trial
* absent consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1900 (Actual)
Dates: Start 2005-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
to compare the rate of fetal extractions between a systematic practice of an echography of presentation and the vaginal touch only one usually realized during the labor. | TWO DAYS
  to compare the rate of fetal extractions between a systematic practice of an echography of presentation and the vaginal touch only one usually realized during the labor.

SECONDARY OUTCOMES:
to optimize the coverage delivery in case of extraction by pair of forceps or suction cup. | two days
  If systematic echography during labor optimize the coverage delivery in case of extraction by pair of forceps or suction cup.

CONTACTS AND LOCATIONS:
Overall Officials: patrick Rozenberg, PU-PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Chi Poissy St Germain, Poissy, France